CLINICAL TRIAL: NCT00116272
Title: OTIS Autoimmune Diseases in Pregnancy Project
Brief Title: Organization of Teratology Information Services (OTIS) Autoimmune Diseases in Pregnancy Project
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20040246; NCT01017016 (obsolete NCT alias)
Record Dates: First submitted 2005-06-28; First posted 2005-06-29 (Estimated); Results first posted 2015-09-21 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2015-08

CONDITIONS: Pregnancy
Keywords: pregnancy; Autoimmune Disease
MeSH Terms: conditions — Autoimmune Diseases | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: None Retained — This is a prospective & observational, exposure cohort study
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Etanercept-Exposed: Pregnant women with a current diagnosis of rheumatoid arthritis (RA), juvenile rheumatoid arthritis (JRA), ankylosing spondylitis (AS), psoriatic arthritis (PsoA) or psoriasis (PsO) who used etanercept in the first trimester of pregnancy for any length of time.
  Interventions: Drug: Etanercept
- Diseased Controls: Pregnant women with a current diagnosis of RA, JRA, AS, PsA, or PsO who did not use etanercept or any tumor necrosis factor (TNF) antagonist during pregnancy.
- Non-Diseased Historical Comparison: Pregnant women not diagnosed with RA, JRA, AS, PsoA, or PsO who did not use etanercept or any TNF antagonist at any time in pregnancy and were not exposed to any known human teratogen during pregnancy. This cohort consists of historical controls enrolled in other pregnancy outcome studies selected to match pregnant women in the exposed cohort.

INTERVENTIONS:
Drug: Etanercept — Pregnant women previously exposed to etanercept during the first trimester. Etanercept was not administered in this non-interventional study.
  Other Names: Enbrel
  Groups: Etanercept-Exposed

SUMMARY:
The purpose of the study is to evaluate the effect of etanercept when used in the first trimester of pregnancy with respect to major structural birth defects of newborns. This is an observational study only - no investigational product is used.

DETAILED DESCRIPTION:
This pregnancy registry cohort study will be conducted by the Organization of Teratology Information Specialists (OTIS) which is a network of university and health department based telephone information centers serving pregnant women and health care providers throughout North America.

Participants in the first two cohorts are recruited concurrently from callers to OTIS centers, from health care providers and through direct to consumer marketing efforts. The source of historical controls is archived data on pregnancies that have been followed through the California Teratogen Information Service's Clinical Research Program located at the University of California San Diego.

ELIGIBILITY:
Cohort 1 Inclusion Criteria: Eligible subjects will be currently pregnant women residing in the US or Canada who have had any exposure to etanercept for treatment of Rheumatoid Arthritis (RA), Juvenile RA, Ankylosing Spondylitis (AS), Psoriatic Arthritis (PsoA) or Psoriasis (PsO) at any time during the first trimester of pregnancy which is defined as the period between first day of the last menstrual period (i.e., within two weeks of conception) up to and including the 12th week after the first day of the last menstrual period (LMP) - Eligible subjects must have documentation of an exposure to etanercept during the first trimester of pregnancy.

Cohort 2 Inclusion Criteria: Eligible subjects will be currently pregnant women residing in the US or Canada who have not taken etanercept or any TNF antagonist for treatment of RA, JRA, AS, PsoA or PsO at any time in the current pregnancy or within two months prior to the first day of the last menstrual period (LMP).

Cohort 3 Inclusion Criteria: Eligible subjects will be pregnant women who were residing in the US or Canada who had not been diagnosed with RA, JRA, AS, PsoA or PsO and had not been exposed to a known human teratogen during the index pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort 1: Exposure Cohort (300 subjects) Cohort 2: Matched diseased control Cohort (300 subjects) Cohort 3: Non-diseased Control Cohort (300 subjects)
Sampling Method: Non-Probability Sample
Enrollment: 830 (Actual)
Dates: Start 2005-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Research Site, San Diego, California, United States

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited concurrently from callers to Organization of Teratology Information Specialists (OTIS) centers, from health care providers and through direct to consumer marketing efforts.
  A third cohort of historical controls including 296 women was also included in the study but are not included in the results of this report.
Pre-assignment Details: The first participant was recruited in April, 2005 and recruitment continued through March 19, 2012.
Period: Overall Study
Arm/Group | Etanercept-Exposed | Diseased Controls
Started | 370 | 164
Completed | 359 (Indicates participants with a known outcome of pregnancy) | 158 (Indicates participants with a known outcome of pregnancy)
Not Completed | 11 | 6
Not completed — Lost to Follow-up | 11 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept-Exposed | Diseased Controls | Total
Number analyzed (Participants) | 370 | 164 | 534
Age, Customized [Number; unit: participants] — Maternal Age at Estimated Due Date
  participants
    < 25 years | 21 | 7 | 28
    25 - 29 years | 81 | 34 | 115
    30 - 34 years | 132 | 48 | 180
    > 34 years | 136 | 75 | 211
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 370 | 164 | 534
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic White | 292 | 138 | 430
  Black | 14 | 3 | 17
  Hispanic | 42 | 13 | 55
  Asian/Pacific Islander | 18 | 6 | 24
  Native American | 3 | 4 | 7
  Other | 1 | 0 | 1
Maternal Education [Number; unit: participants]
  < 12 years | 9 | 4 | 13
  12 - 15 years | 118 | 42 | 160
  > 15 years | 243 | 118 | 361
Hollingshead Socioeconomic Category [Number; unit: participants] — Based on four-factor Hollingshead categories incorporating maternal and paternal education and occupation; highest socioeconomic status category = 1; lowest socioeconomic status category = 5.
  participants
    1 | 134 | 69 | 203
    2 | 145 | 67 | 212
    3 | 59 | 19 | 78
    4 | 23 | 6 | 29
    5 | 7 | 3 | 10
    Missing | 2 | 0 | 2
Pre-pregnancy Height [Mean (Standard Deviation); unit: cm] | 164.7 (7.1) | 166.7 (7.0) | 165.3 (7.1)
Pre-pregnancy Body Weight [Mean (Standard Deviation); unit: kg] | 70.2 (18.14) | 68.3 (16.5) | 69.6 (17.8)
Gravidity Category [Number; unit: participants]
  1 pregnancy | 135 | 62 | 197
  2 -3 pregnancies | 163 | 78 | 241
  4 -5 pregnancies | 60 | 21 | 81
  ≥ 6 pregnancies | 12 | 3 | 15
Parity Category [Number; unit: participants]
  0 births | 193 | 88 | 281
  1 -2 births | 153 | 69 | 222
  3 - 4 births | 22 | 7 | 29
  ≥ 5 births | 2 | 0 | 2
Previous Spontaneous Abortion [Number; unit: participants]
  0 | 265 | 117 | 382
  1 | 73 | 30 | 103
  2 | 22 | 11 | 33
  ≥ 3 | 10 | 6 | 16
Previous Elective Terminations [Number; unit: participants]
  0 | 314 | 150 | 464
  1 | 49 | 12 | 61
  2 | 5 | 1 | 6
  ≥ 3 | 2 | 1 | 3
Previous Preterm Delivery [Number; unit: participants]
  Yes | 37 | 6 | 43
  No | 333 | 158 | 491
Any Previous Child with Birth Defect [Number; unit: participants]
  Yes | 20 | 8 | 28
  No | 350 | 156 | 506
In Vitro Fertilization (IVF) with This Pregnancy [Number; unit: participants]
  Yes | 27 | 5 | 32
  No | 343 | 159 | 502
Gestational Age at Time of Enrollment [Number; unit: participants]
  < 13 weeks | 196 | 84 | 280
  13 - 19.9 weeks | 99 | 58 | 157
  ≥ 20 weeks | 75 | 22 | 97
Referral Source Category [Number; unit: participants]
  Sponsor | 37 | 1 | 38
  Health-care Professional (HCP) | 185 | 53 | 238
  Internet | 65 | 27 | 92
  Patient Support Group | 0 | 4 | 4
  OTIS Member Service | 29 | 69 | 98
  Other | 53 | 10 | 63
  Missing | 1 | 0 | 1
Geographic Area of Residence [Number; unit: participants]
  United States | 338 | 136 | 474
  Canada | 31 | 27 | 58
  Missing | 1 | 1 | 2
Maternal Comorbidities [Number; unit: participants] — Participants could have more than one comorbidity
  participants
    Thyroid Disease | 45 | 23 | 68
    Asthma | 48 | 33 | 81
    Other Autoimmune Disease | 43 | 17 | 60
    Antidepressant Medication Use in Any Trimester | 28 | 14 | 42
    Pre-gestational Hypertension | 19 | 10 | 29
    Preeclampsia | 11 | 8 | 19
    Other Psychiatric Conditions | 64 | 32 | 96
    Infections | 274 | 114 | 388
Prenatal Multivitamin or Folic Acid Supplements [Number; unit: participants]
  Began Prior to Conception | 217 | 114 | 331
  Post-conception Only | 148 | 50 | 198
  Not Taken at All | 5 | 0 | 5
Alcohol Use During Pregnancy [Number; unit: participants]
  Yes | 177 | 80 | 257
  No | 193 | 84 | 277
Tobacco Use During Pregnancy [Number; unit: participants]
  Yes | 40 | 17 | 57
  No | 330 | 147 | 477
Major Known or Suspected Human Teratogens [Number; unit: participants]
  Yes | 14 | 11 | 25
  No | 356 | 153 | 509
Intended Pregnancy [Number; unit: participants]
  Yes | 264 | 123 | 387
  No | 106 | 41 | 147
Primary Disease (RA, JRA, PsA or AS) [Number; unit: participants]
  Yes | 311 | 117 | 428
  No | 59 | 47 | 106
Duration of Disease [Mean (Standard Deviation); unit: years] — Year was known, but month and date were not known for all cases, therefore Jan 1 of the year of diagnosis through the 1st day of the last menstrual period for the index pregnancy was used to calculate duration of disease. In cases where the woman had multiple study diseases, the earliest known year of the "primary disease" diagnosis was used to calculate duration. Five participants in the Etanercept-Exposed Group were missing year of diagnosis.
  years | 9.8 (7.9) | 10.0 (9.1) | 9.9 (8.3)
Prednisone and/or Systemic Oral Corticosteroid [Number; unit: participants]
  Yes | 163 | 65 | 228
  No | 207 | 99 | 306
Disease Severity Score - RA [Mean (Standard Deviation); unit: units on a scale] — RA1 disease severity score expressed as the Health Assessment Questionnaire-Disability Index (HAQ-DI) summary score; possible score ranges from 0-3 with higher score representing higher severity/disability.
  RA1 disease severity score at intake missing for 2 participants in the Etanercept-Exposed Group and 1 participant in the Diseased Controls Group.
  units on a scale | 0.5 (0.6) | 0.6 (0.6) | 0.5 (0.6)
Disease Severity Score - PsO [Mean (Standard Deviation); unit: units on a scale] — Maternal rating of overall severity of psoriasis measured using Global Assessment of Psoriasis, possible score 0-5 with higher score indicating more severe disease.
  units on a scale | 2.0 (1.5) | 1.9 (1.1) | 1.9 (1.4)
Exposed to Etanercept [Number; unit: participants] — the first trimester of pregnancy is defined as the period between the estimated date of conception (DOC) to the 11th week post-conception. The date of conception is defined as 14 days prior to the next expected menstrual period.
  participants
    First Trimester | 344 | 0 | 344
    Last Menstrual Period to Date of Conception | 8 | 0 | 8
    2nd and/or 3rd Trimester Only | 13 | 0 | 13
    Started Prior to DOC, End Date Unavailable | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Infants With Major Birth Defects in Pregnancies Ending With Live-born Infants
Description: A major structural defect is defined as a defect which has either cosmetic or functional significance to the child (e.g., a cleft lip). The Registry used the Metropolitan Atlanta Congenital Defects Program (MACDP) birth defect classification system, with some specified modifications that are appropriate for cohort studies as opposed to case-control studies.
Time Frame: From birth through 1 year of age
Population: Includes multiple pregnancies ending in at least 1 live-born infant; any 1 or more malformed live-born infants counted as 1 major malformation outcome in the numerator, and 1 pregnancy outcome in the denominator. Only women exposed to etanercept in the 1st trimester are included in the Etanercept-Exposed cohort.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 319 | 144
percentage of participants | 9.4 | 3.5
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Odds Ratio (OR) = 2.77, 95% CI 2-sided [1.04 to 7.35] — Adjusted oddds ratio for major structural defects in women exposed to etanercept in their 1st trimester versus not exposed computed using logistic regression adjusted for propensity score comprised of asthma and maternal height

2. Primary Outcome: Percentage of Infants With Major Birth Defects in All Pregnancies
Description: as for outcome 1
Time Frame: From birth through 1 year of age
Population: Includes multiple pregnancies counted as 1 outcome; any 1 or more malformed infant counted as 1 major malformation in the numerator and 1 outcome in the denominator. Excludes 9 lost-to-follow-up in Etanercept-Exposed and 6 in Diseased Controls cohort. Only women exposed to etanercept in 1st trimester are included in the Etanercept-Exposed cohort.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 335 | 158
percentage of participants | 9.9 | 4.4
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Odds Ratio (OR) = 2.37, 95% CI 2-sided [1.02 to 5.52] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Infants With Any 3 or More Minor Birth Defects
Description: A minor structural defect is defined as a defect which occurs in less than 4 percent of the population but which has neither cosmetic nor functional significance to the child (e.g., complete 2,3 syndactyly of the toes). The Registry used the Metropolitan Atlanta Congenital Defects Program (MACDP) birth defect classification system, with some specified modifications that are appropriate for cohort studies as opposed to case-control studies.
Time Frame: From birth through 1 year of age
Population: Children born to enrolled participants during the study who received the dysmorphological exam. Includes singletons and 1 randomly selected twin from twin pairs. Only women exposed to etanercept in the 1st trimester are included in the Etanercept-Exposed cohort.
Measure: Number; unit: percentage of infants
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 257 | 111
percentage of infants | 25.7 | 22.5
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.70 to 2.01] — Unadjusted Odds Ratio computed using logistic regression. No adjusted estimate was computed due to no confirmed confounder

4. Secondary Outcome: Percentage of Infants With a Specific Pattern of Any 3 or More Minor Birth Defects
Description: A minor structural defect is defined as a defect which occurs in less than 4 percent of the population but which has neither cosmetic nor functional significance to the child (e.g., complete 2,3 syndactyly of the toes). A pattern is defined as at least the same 3 specific minor malformations occurring in at least two infants in the exposed group.
Time Frame: From birth through 1 year of age
Population: Children born to enrolled participants who received the dysmorphological exam. Includes multiples who received the exam for consideration of pattern; co-twins with the same 3 or more minor defects could not constitute a pattern on their own. Only women exposed to etanercept in the 1st trimester are included in the Etanercept-Exposed cohort.
Measure: Number; unit: percentage of infants
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 262 | 113
percentage of infants | 2.3 | 0.0

5. Secondary Outcome: Percentage of Pregnancies Ending in Spontaneous Abortion
Description: Computed using Kaplan-Meier estimate at 20 weeks gestation, accounting for left truncation due to varying time in gestation at enrollment. In multiple pregnancies ending in at least 1 live-born infant, the live birth outcome is included in the analysis. In multiples ending in no live birth outcomes, the spontaneous abortion is counted as 1 event.
Time Frame: 9 months
Population: Participants enrolled and exposed to etanercept prior to 20 weeks gestation (Etanercept-Exposed) or enrolled prior to 20 weeks gestation (Diseased Controls).
Measure: Number (95% Confidence Interval); unit: percentage of pregnancies
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 288 | 137
percentage of pregnancies | 14.7 [7.4 to 28.3] | 28.8 [16.0 to 48.5]
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.20 to 1.12] — Adjusted HR computed using Cox proportional hazards regression adjusted for propensity score comprised of referral source (3 categories: OTIS, Pharmaceutical Company/Sponsor/HCP, Patient Support Group/Internet/Other), and maternal height

6. Secondary Outcome: Percentage of Participants With Pre-term Delivery
Description: A pretem delivery is defined as prior to 37 weeks gestation. Computed using Kaplan-Meier estimate at 37 weeks' gestation, accounting for left truncation due to varying time in gestation at enrollment. Multiple births are excluded.
Time Frame: 9 months
Population: Participants enrolled and exposed to etanercept prior to 37 weeks gestation (Etanercept-Exposed) or enrolled prior to 37 weeks gestation (Diseased Controls), and excluding multiple births.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 324 | 142
percentage of participants | 13.9 [10.5 to 18.2] | 10.0 [6.1 to 16.3]
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Hazard Ratio (HR) = 1.60, 95% CI 2-sided [0.86 to 2.98] — Adjusted HR computed using Cox proportional hazards regression adjusted for preeclampsia

7. Secondary Outcome: Gestational Age at Delivery (GAD) of Live Births
Time Frame: At birth
Population: Live births in women enrolled and exposed to etanercept prior to 37 weeks' gestation (Etanercept-Exposed) or enrolled prior to 37 weeks gestation (Diseased Controls), excluding multiple births.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 324 | 142
weeks | 38.6 (2.2) | 38.8 (2.0)
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Adjusted Difference = -0.20, 95% CI 2-sided [-0.65 to 0.26] — Computed using linear regression, directly adjusted for referral source (not collapsed), vitamin use (not collapsed), preeclampsia, and asthma because propensity score adjustment was not balanced

8. Secondary Outcome: Birth Weight Among Full Term Infants
Time Frame: At birth
Population: Live birth full-term infants, excluding multiple births, where data were available
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 282 | 128
g | 3399.1 (434.9) | 3380.2 (447.0)
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Adjusted Difference = 21.79, 95% CI 2-sided [-83.32 to 126.91] — Computed using linear regression, directly adjusted for asthma, RA2 severity score at 32 weeks, and disease severity score imputation indicator because propensity score adjustment was not balanced

9. Secondary Outcome: Birth Length Among Full Term Infants
Time Frame: At birth
Population: Live birth full-term infants, excluding multiple births, where data were available
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 277 | 127
cm | 50.8 (2.6) | 50.7 (2.4)
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Adjusted Difference = 0.10, 95% CI 2-sided [-0.44 to 0.63] — Computed using linear regression, adjusted for propensity score comprised of preeclampsia and asthma

10. Secondary Outcome: Birth Head Circumference Among Full Term Infants
Time Frame: At birth
Population: Live birth full-term infants, excluding multiple births, where data were available
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 253 | 116
cm | 34.4 (1.6) | 34.5 (1.5)
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Adjusted Difference = -0.09, 95% CI 2-sided [-0.43 to 0.26] — Computed using linear regression, adjusted for maternal age (categorical)

11. Secondary Outcome: Percentage of Infants With Small for Gestational Age Birth Weight
Description: Small for gestational age is defined as ≤ 10th percentile for sex and gestational age using National Center for Health Statistics (NCHS) / Center for Disease Control (CDC) growth curves.
Time Frame: At birth
Population: Live-born infants, excluding multiple births, where data were available.
Measure: Number; unit: percentage of infants
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 324 | 141
percentage of infants | 6.8 | 10.6
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.22 to 1.05] — Computed using logistic regression, adjusted for propensity score comprised of maternal height, referral source (OTIS, Sponsor/HCP, Patient Support Group/Internet/Other), PsO disease severity score at 32 weeks, & disease severity imputation indicator

12. Secondary Outcome: Percentage of Infants With Small for Gestational Age Birth Length
Description: as for outcome 11
Time Frame: At birth
Population: Live-born infants, excluding multiple births, where data were available.
Measure: Number; unit: percentage of infants
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 317 | 139
percentage of infants | 4.7 | 6.5
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.31 to 1.68] — Unadjusted Odds Ratio computed using logistic regression. An adjusted estimate was not computed due to the small number of events

13. Secondary Outcome: Percentage of Infants With Small for Gestational Age Birth Head Circumference
Description: as for outcome 11
Time Frame: At birth
Population: Live-born infants, excluding multiple births, where data were available.
Measure: Number; unit: percentage of infants
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 287 | 125
percentage of infants | 17.1 | 14.4
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.40 to 1.57] — [estimate comment as in outcome 11, analysis 1]

14. Secondary Outcome: Postnatal Weight Percentile at One Year
Time Frame: 1 year after birth
Population: Live-born infants, excluding multiple births, where 1-year data were available
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 248 | 108
percentile | 45.1 (30.1) | 44.1 (28.6)
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Adjusted Difference = 0.20, 95% CI 2-sided [-7.59 to 7.99] — Computed using linear regression, adjusted for propensity score comprised of maternal height, vitamin use, primary disease, RA disease severity score at 32 weeks, PsO disease severity score at intake & 32 weeks, disease severity imputation indicators

15. Secondary Outcome: Postnatal Length Percentile at One Year
Time Frame: 1 year after birth
Population: Live-born infants, excluding multiple births, where 1-year data were available
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 251 | 110
percentile | 60.1 (29.7) | 62.3 (27.9)
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Adjusted Difference = 1.53, 95% CI 2-sided [-5.76 to 8.81] — Computed using linear regression, adjusted for propensity score comprised of maternal height, maternal age (categorical), and referral source (3 categories: OTIS, Pharmaceutical Company/Sponsor/HCP, Patient Support Group/Internet/Other)

16. Secondary Outcome: Postnatal Head Circumference Percentile at One Year
Time Frame: 1 year after birth
Population: Live-born infants, excluding multiple births, where 1-year data were available
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 243 | 108
percentile | 63.9 (28.3) | 63.8 (27.0)
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Adjusted Difference = 0.27, 95% CI 2-sided [-6.12 to 6.65] — Computed using linear regression. Directly adjusted for infant sex and other autoimmune diseases because propensity score adjustment was not balanced

17. Secondary Outcome: Percentage of Infants at One Year of Age With Small for Gestational Age Weight
Description: Postnatal growth deficiency defined as ≤ 10th centile for chronological age. Age adjusted for gestational age at delivery if child was less than 12 months of age at postnatal measurement, unadjusted if ≥ 12 months of age at postnatal measurement.
Time Frame: 1 year after birth
Population: Live-born infants, excluding multiple births, where data were available.
Measure: Number; unit: percentage of infants
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 248 | 108
percentage of infants | 14.5 | 13.9
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.37 to 1.62] — Computed using logistic regression, adjusted for propensity score comprised of maternal height, RA disease severity score at 32 weeks, and disease severity score imputation indicator

18. Secondary Outcome: Percentage of Infants at One Year of Age With Small for Gestational Age Length
Description: as for outcome 17
Time Frame: 1 year after birth
Population: Live-born infants, excluding multiple births, where data were available.
Measure: Number; unit: percentage of infants
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 251 | 110
percentage of infants | 7.2 | 5.5
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.43 to 3.14] — Computed using logistic regression, adjusted for propensity score comprised of country (U.S., Canada), primary disease, and maternal height

19. Secondary Outcome: Percentage of Infants at One Year of Age With Small for Gestational Age Head Circumference
Description: as for outcome 17
Time Frame: 1 year after birth
Population: Live-born infants, excluding multiple births, where data were available.
Measure: Number; unit: percentage of infants
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 243 | 108
percentage of infants | 4.1 | 4.6
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.29 to 2.65] — [estimate comment as in outcome 12, analysis 1]

20. Secondary Outcome: Percentage of Infants With Reported Serious or Opportunistic Infections Through One Year
Time Frame: From birth to 1 year
Population: Live-born infants, including singletons and 1 randomly selected twin from multiple pregnancies, born to enrolled women exposed to etanercept at any time during pregnancy (Etanercept-Exposed).
Measure: Number; unit: Percentage of infants
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 342 | 144
Percentage of infants | 5.3 | 4.2
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.47 to 4.02] — Unadjusted Odds Ratio computed using logistic regression. An adjusted estimate was not computed due to no confirmed confounder

21. Secondary Outcome: Percentage of Infants Diagnosed With Any Malignancy Through One Year of Age
Time Frame: From birth to 1 year
Population: as for outcome 20
Measure: Number; unit: Percentage of infants
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 342 | 144
Percentage of infants | 0 | 0

22. Secondary Outcome: Percentage of Infants With Abnormal Results on Ages and Stages Questionnaire (ASQ)
Description: The ASQ-3 evaluates 5 domains of development: communication, gross motor, fine motor, problem solving, and personal-social. Each domain has a set of 6 items and parents rate the most appropriate answer for the presence of each skill: "Yes," "Sometimes," "Not Yet," with point values of 10, 5, or 0, respectively. Each domain question set is totaled independently and compared against statistically derived cutoffs that are set at 2 standard deviations below the mean. The percentage of infants below the cut-off or close to the cutoff (borderline) is reported.
Time Frame: 1 year after birth
Population: Live-born infants, including singletons and 1 randomly selected twin from multiple pregnancies, where data were available.
Measure: Number; unit: Percentage of infants
Arm/Group | Etanercept-Exposed | Diseased Controls
Number analyzed (Participants) | 287 | 117
Percentage of infants | 28.2 | 27.4
Statistical Analysis 1: Comparison: Etanercept-Exposed vs Diseased Controls; Test type: Superiority or Other; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.65 to 1.69] — [estimate comment as in outcome 20, analysis 1]

ADVERSE EVENTS:
Time Frame: Mothers (enrolled women) were assessed during pregnancy (up to 9 months) and up to 6 weeks after delivery; Infants were assessed for up to 1 year after birth.
Description: Only Serious Adverse Events were collected for this study.
Groups:
- Mothers Diseased Control: Pregnant women with a current diagnosis of RA, JRA, AS, PsA, or PsO who did not use etanercept or any tumor necrosis factor (TNF) antagonist during pregnancy.
- Mothers Etanercept Exposed: Pregnant women with a current diagnosis of rheumatoid arthritis (RA), juvenile rheumatoid arthritis (JRA), ankylosing spondylitis (AS), psoriatic arthritis (PsoA) or psoriasis (PsO) who used etanercept in the first trimester of pregnancy for any length of time.
- Infants Diseased Control: Infants born to pregnant women with a current diagnosis of RA, JRA, AS, PsA, or PsO who did not use etanercept or any tumor necrosis factor (TNF) antagonist during pregnancy.
- Infants Etanercept Exposed: Infants born to pregnant women with a current diagnosis of rheumatoid arthritis (RA), juvenile rheumatoid arthritis (JRA), ankylosing spondylitis (AS), psoriatic arthritis (PsoA) or psoriasis (PsO) who used etanercept in the first trimester of pregnancy for any length of time.
Arm/Group | Mothers Diseased Control | Mothers Etanercept Exposed | Infants Diseased Control | Infants Etanercept Exposed
Serious Adverse Events (participants affected / at risk) | 18/164 | 37/370 | 12/146 | 59/352
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mothers Diseased Control (N=164) | Mothers Etanercept Exposed (N=370) | Infants Diseased Control (N=146) | Infants Etanercept Exposed (N=352)
Neutropenia neonatal (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Atrial hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 1
Pulmonary valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 2
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 9
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Cleft palate (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Congenital aortic valve incompetence (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Congenital cardiovascular anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 2
Congenital cystic lung (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Congenital eye disorder (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Congenital gastric anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 2
Congenital mitral valve incompetence (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 2
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Double ureter (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Epispadias (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Haemangioma congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Heart block congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Hypospadias (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Kidney duplex (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Limb reduction defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Microcephaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 3
Micropenis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Neurofibromatosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Noonan syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 2
Polydactyly (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Pulmonary artery stenosis congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 2
Pulmonary valve stenosis congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 4
Transposition of the great vessels (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Trisomy 13 (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Trisomy 21 (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 1
Turner's syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 2
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 3
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Necrotising colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 1 | 0 | 1
Developmental delay (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 2 | 0 | 0
Group B streptococcus neonatal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 1 | 0 | 1
Meningitis neonatal (Infections and infestations) | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 2 | 1 | 7
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 2
Pyelonephritis (Infections and infestations) | 1 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 3
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis neonatal (Infections and infestations) | 0 | 0 | 0 | 6
Septic shock (Infections and infestations) | 0 | 0 | 0 | 2
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Uterine infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Blood glucose abnormal (Investigations) | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 13 | 17 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 3
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Reflux nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1
Shortened cervix (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bronchomalacia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Immature respiratory system (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary artery stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Abortion induced (Surgical and medical procedures) | 1 | 3 | 0 | 0
Transplant (Surgical and medical procedures) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.